CLINICAL TRIAL: NCT04997460
Title: Diabetes Type One in Pregnancy and Continuous Glucose Monitoring - Observational Prospective Study in Croatia
Brief Title: Diabetes Type One in Pregnancy and Continuos Glucose Monitoring
Acronym: DIP1/CRO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Gloria Leksic, Resident, Clinical Hospital Centre Zagreb
Other Study IDs: 8.1-21/4-2, 02/21 AG
Record Dates: First submitted 2021-07-06; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Large-for-gestational-age Neonates; Glycemic Variability; Hypoglycemia; Pregnancy Outcomes; C-peptide
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Type I diabetes mellitus (T1DM) affects about 0.1-0.2% of all pregnancies. T1DM in pregnancy increases the risk of maternal and neonatal complications.

Continuous glucose monitoring systems (CGM) provide a continuous display of measured glucose. Studies have shown improved pregnancy outcomes for patients with T1DM using CGM when compared to capillary blood glucose measurements.

This prospective observational study analyses impact of glycemic variability on development of large-for-gestational-age neonates and effects of hypoglycemia during pregnancy on pregnancy outcomes.

Furthermore, overall glycemic regulation, different insulin metrics and C-peptide concentration during pregnancy will also be assesed.

DETAILED DESCRIPTION:
Up to 200 patients with type one diabetes will be enrolled in the study during first trimester of pregnancy. Medical history, clinical examination, anthropometric measurements and laboratory work-up will be obtained at first visit. Glucose metrics are provided from continuous glucose monitoring systems and blood glucose measurements .

Following the initial evaluation, patients will be regularly examined in the hospital setting once a month during pregnancy. Following evaluations will include the same procedures as the first one.

Pregnancy outcomes that will be analysed: spontaneous abortion, preterm birth, large-for-gestational-age neonates, macrosomia, small-for-gestational-age neonates, birth weight, congenital anomalies, APGAR score, neonatal hypoglycemia, intensive care unit admission for mother and/or infant.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of type one diabetes
* duration of the disease for minimum of one year before inclusion in the study
* multiple daily insulin injection therapy or insulin pump
* glycemia monitoring with continuous glucose monitoring systems (FreeStyle Libre Flash Glucose Monitoring System, Abott) for a minimum of 3 months before inclusion in the study
* glucose data availability from the sensor > 80% for a determined period of monitoring
* patient age > 18 years and < 40 years
* available medical records from the preconception period (3 months before conception)
* first trimester of pregnancy
* body mass index < 25kg/m2
* glycated haemoglobin < 7.0%
* signed informed consent

Exclusion Criteria:

* other types of diabetes except type one: type 2 diabetes, diabetes developed during pregnancy, diabetes as a result of genetic defect of beta-cells of the pancreas
* using other therapy besides insulin in treating diabetes
* changes to the specific insulin therapy in preconception period or during pregnancy; defined as switching from multiple daily insulin injection therapy to insulin pumps and vice versa
* patient's inability for regular hospital visits (defined as once monthly during pregnancy)
* patients unable to understand the protocol and the goal of the study
* patients unable to read and write
* multiple pregnancy
* glycated haemoglobin > 7.0% in all pregnancy trimesters
* significant weight gain during pregnancy (>20 kilograms)
* glucose data availability from the sensor < 80%
* unavailability of preconception medical records
* unavailability of medical records from pregnancy and pregnancy outcomes

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Patients enrolled in the study are women who are patients of the Clinic for gynecology and obstetrics and who match the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2024-01-11 (Estimated); Study Completion 2024-01-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of large-for-gestational-age neonates | 9 months
  Incidence of large-for-gestational-age neonates will be determined in group of patients with increased glycemic variability (%CV> 36%) and in the group of patients with normal glycemic variability (%CV < 36%) during different pregnancy trimesters.
  Glycemic variability parameters are available from continuous glucose monitoring system:percent coefficient of variation (%CV), interquartile range (IQR), standard deviation (SD).
Correlation of glycated hemoglobin and glycemic variability | 9 months
  Correlation of glycemic variability parameters (%CV, IQR, SD) and glycated hemoglobin in different pregnancy trimesters will be performed.Both parameters are available from continuos glucose monitoring systems.

SECONDARY OUTCOMES:
Pregnancy outcomes - maternal and fetal | 9 months
  Effects of hypoglycemia on pregnancy outcomes will be analysed. Pregnancy outcomes included in the analysis: spontaneous abortion, preterm birth, large-for-gestational-age neonates, macrosomia, small-for-gestational-age neonates, birth weight, congenital anomalies, APGAR score, neonatal hypoglycemia, intensive care unit admission for mother and/or infant.
  Hypoglycemia will be assesed through parameters available from continuos glucose monitoring systems (low glucose events, time spent below target).
Correlation of hypoglycemia and glycemic variability | 9 months
  Correlation between hypoglycemia parameters (time below target, low glucose events) and glycemic variability parameters (%CV, SD, IQR) will be performed. Both parameters are available from continuous glucose monitoring systems.

OTHER OUTCOMES:
C-peptide concentration in different pregnancy trimesters | 9 months
  C-peptide concentration will be determined from venous blood sample in every pregnancy trimester.

CONTACTS AND LOCATIONS:
Overall Officials: Maja Baretic, Study Director — Clinical Hospital Centre Zagreb; Marina Ivanisevic, Study Chair — Clinical Hospital Centre Zagreb; Gloria Leksic, Principal Investigator — Clinical Hospital Centre Zagreb
Locations (1):
- University hospital centre Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Undecided